CLINICAL TRIAL: NCT04873505
Title: Functional Validation of Lactobacillus Containing Oral Tablet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A-BR-109-047
Record Dates: First submitted 2021-04-22; First posted 2021-05-05 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Periodontal Disease
Keywords: Caries; Periodontal disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Troches (Experimental): 25 persons take one probiotic troche after each meal.
  Interventions: Dietary Supplement: troches
- Troches do not contain probiotics (Placebo Comparator): 25 persons take one troche that does not contain probiotics after each meal.
  Interventions: Dietary Supplement: troches

INTERVENTIONS:
Dietary Supplement: troches — Take one troche after each meal.

SUMMARY:
Dental caries and periodontal disease are the two most common diseases in dentistry. Caries was caused by the acidic environment produced through the interaction of oral flora (biofilm) and fermentable food residues on the tooth surface over time thus to destroying the tooth structure. Periodontal disease was also highly associated with microorganisms in the periodontal tissues and the inflammatory response of the host that irritate and destruct periodontal and bone tissues. Recent studies have found that both stress and eating habits are associated with decline in oral health. Probiotics have been traditionally used for prevention and treatment of gastrointestinal diseases. In the past decade, accumulated studies further indicate that imbalance of oral microflora is highly related to oral diseases thus probiotics has been suggested for maintaining oral health. It is thus conceivable that probiotics as a buccal tablet may potentially restore the balance of oral flora providing a novel strategy to combat oral diseases. Such strategy may also harbor great opportunities for the long-term management of dental caries and periodontal infections. In order to evaluate the efficacy of probiotics buccal tablet in rebalancing oral flora and control to reduce the incidence of dental caries and periodontal diseases, the investigators aimed to conduct a comprehensive clinical trials for subsequent product optimization.

Grape King Biotechnology Co., Ltd. has successfully developed oral tablet mainly composed of Lactobacillus plantarum GKD7 and Pediococcus acidilactici GKA4. These two probiotics were found to inhibit caries through producing protective biofilms thus are more effective than commercially available anti-tooth decay products. To evaluate the future potential of clinical applications of the related products series and the impact on oral health-related indicators, the investigators will explore the changes in the the following disease associated indexes before and after using the oral tablet. These include periodontal pocket depth, the gingival inflammation index, the plaque index, and the ratio of Firmicutes, Bacteroidetes, Streptococcus mutans, and Porphyromonas gigivalis, as well as quantification of total bacteria. This clinical study will be performed in Department of Stomatology in NCKUH in collaboration with periodontics session and Family Dentistry session. A total of 50 healthy individuals within the range of 20~65 years old will be enrolled.

DETAILED DESCRIPTION:
The following parameters will be collected and analyzed: periodontal pocket depth, the gingival inflammation index, the plaque index, and the ratio of Firmicutes/ Bacteroidetes/Streptococcus mutans/Porphyromonas gigivalis, as well as total count of microorganisms from the plaque collected.

ELIGIBILITY:
Inclusion Criteria:

* 20~65 years old
* At least 20 teeth except wisdom teeth

Exclusion Criteria:

* Smoking habits
* Oral cancer or other serious oral diseases.
* Pregnancy
* Severe chronic diseases
* Coagulation diseases
* Long-term or regular use of medication (anti-epileptics, antihistamines, anti-inflammatory, sedatives, tranquilizers, analgesics, Chinese herbs)
* Allergy to test products

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Periodontal pocket depth | 1 hour
  The probe should be walked around each tooth, and the probing depth of each tooth will be recorded in its six aspect (MB, M, DB, ML, L, DL)

SECONDARY OUTCOMES:
Gingival index | 30 minutes
  The scores from the six areas of the tooth may be added and divided by six to give the GI for the tooth.
  By adding the indices for the teeth and dividing by the total number of teeth examined, the Gl for the individual is obtained.
Plaque index | 1 hour
  The disclosing solution is painted on all exposed tooth surfaces. After the patient has rinsed, the operator, using an explorer or the tip of a probe, examines each stained surface for soft accumulations at the dentogingival junction. When found, they are recorded by making a dash in the appropriate spaces on the record form.Silmilar to the gingival index, each of the six gingival areas of the tooth will be examined and recorded.
  The overall plaque index is calculated by dividing the number of plaque containing surfaces with the total number of available surfaces.
Plaque microorganisms | 30 minutes
  The ratio of Firmicutes/ Bacteroidetes/Streptococcus mutans/Porphyromonas gigivalis, as well as total count of microorganisms from the plaque collected.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Ying Chang, Study Chair — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No